CLINICAL TRIAL: NCT01692782
Title: A Randomized, Double Blind, Parallel Group, Multicenter Efficacy and Safety Study of SEP-225289 Versus Placebo in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Adult Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP360-201
Record Dates: First submitted 2012-09-18; First posted 2012-09-25 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Adult Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention deficit hyperactivity disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — SEP 225289; 4-(3,4-dichlorophenyl)-1,2,3,4-tetrahydronaphthalen-1-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SEP-225289 4mg (Experimental): SEP-225289 4mg once daily taken as a combination of SEP-225289 2mg and placebo capsules to achieve 4mg QD doses
  Interventions: Drug: SEP-225289
- SEP-225289 8mg (Experimental): SEP-225289 8mg once daily taken as a combination of SEP-225289 2mg and placebo to achieve 8mg QD doses
  Interventions: Drug: SEP-225289
- Placebo (Placebo Comparator): 4 capsules of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP-225289 — SEP-225289 4mg once daily
  Other Names: Dasotraline
  Arms: SEP-225289 4mg
Drug: SEP-225289 — SEP-225289 8mg once daily
  Other Names: Dasotraline
  Arms: SEP-225289 8mg
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
A Phase 2 study of SEP-225289 in adults with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, parallel-group, multicenter, outpatient study evaluating the efficacy and safety of SEP 225289 in adults with ADHD using 2 oral dosages (4 or 8 mg SEP 225289 once daily [QD]) versus placebo over a 4 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets Diagnostic and Statistical Manual of Mental Disorders Fourth Edition; Text Revision (DSM-IV-TR) criteria for a primary diagnosis of ADHD (inattentive, hyperactive, or combined subtype) established by a comprehensive psychiatric evaluation that reviews DSM-IV-TR criteria. Diagnosis is confirmed by Conners' Adult ADHD Diagnostic Interview (CAADID) Part 2.
* Subject currently taking medication (stimulant or nonstimulant) for the control of ADHD symptoms has an ADHD RS-IV score of ≥ 22 at screening.
* Subject currently not taking any medication for the purpose of controlling ADHD symptoms has an ADHD RS-IV score of ≥ 26 at screening.
* Subject has a CGI-S score of ≥ 4 at screening.
* Subject has a lifetime history of treatment with at least one medication for ADHD (stimulant or nonstimulant). Subjects may be either medicated or unmedicated for ADHD at the time of screening (all ADHD medications must be washed out during screening).
* Subject has a negative breath alcohol test and a negative urine drug screen (UDS) for any illicit drug at screening, unless a false positive is suspected, in which case the UDS will be repeated. If the subject has a positive drug screen for ADHD medications (ie, methylphenidate or amphetamine) at screening; the subject must have a negative UDS after a washout period at least 3 days prior to baseline.
* Subject is male or a non-pregnant, non-lactating female.
* Female subjects must have a negative serum pregnancy test at screening; women who are post-menopausal (defined as at least 12 months of spontaneous amenorrhea) and those who have undergone hysterectomy or bilateral oophorectomy will be exempted from the pregnancy test.
* Female subjects of childbearing potential and male subjects with female partners of child-bearing potential must agree to use an effective and medically acceptable form of birth control throughout the study period and for one month (30 days) after study completion. Medically acceptable and effective contraceptives include abstinence, prescription hormonal contraceptives (oral, patch, vaginal ring, implant, or injection), diaphragm with spermicide, intrauterine device (IUD), condom with spermicide, surgical sterilization, or vasectomy. For male subjects adequate contraception is defined as abstinence or continuous use of 2 barrier methods of contraception (eg, spermicidal condom).
* Subject is 18 to 55 years old, inclusive, at the time of informed consent. 11. Subject can read well enough to understand the informed consent form and other subject materials.

Exclusion Criteria:

* Subject has a DSM-IV-TR diagnosis of ADHD not otherwise specified.
* Subject is receiving adequate benefit from current ADHD medication in the opinion of the investigator.
* Subject has an Axis I disorder other than ADHD that has been the primary focus of treatment at any time during the 12 months prior to screening.
* Subject has a past history of, or current presentation consistent with, bipolar disorder (including bipolar I, bipolar II, and bipolar not otherwise specified [NOS]), schizophrenia, schizoaffective disorder, or any other psychotic disorder.
* Subject has a history of drug dependence or substance abuse (excluding nicotine and caffeine) within the 12 months prior to screening, as defined by the DSM-IV-TR criteria.
* Subject has a current Axis II disorder per DSM-IV-TR criteria.
* Subject has a history of epilepsy, seizures (except childhood febrile seizures), unexplained syncope or other unexplained blackouts (except single incident), or head trauma with loss of consciousness lasting more than 5 minutes.
* Subject has a currently active medical condition (other than ADHD) that, in the opinion of the investigator, could interfere with the ability of the subject to participate in the study.
* Subject is currently taking an antidepressant medication (eg, bupropion, selective serotonin reuptake inhibitor [SSRI]/ serotonin norepinephrine reuptake inhibitor [SNRI], monoamine oxidase [MAO] blocker, tricyclic, etc) or St. John's Wort.
* Subject is currently taking or has taken within the previous 6 months an anticonvulsant medication (eg, phenytoin, carbamazepine, lamotrigine, valproic acid, etc); antipsychotic medication; or lithium (any lithium preparation or formulation).
* Subject is currently taking an alpha-2 adrenergic receptor agonist (including clonidine and guanfacine).
* Subject has a Body Mass Index (BMI) less than 18 or greater than 35 kg/m2 (refer to Appendix V)
* Subject answers "yes" to "Suicidal Ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at screening (in the past month). Subjects who answer "yes" to this question must be referred to the Investigator for follow-up evaluation.
* Subject has attempted suicide within 2 years prior to the screening period.
* Subject has history of positive test for Hepatitis B surface antigen or Hepatitis C antibody. Note: Subjects with a history of a positive test for Hepatitis B surface antigen or Hepatitis C antibody may be enrolled in the study if they have liver function test results at screening within the normal range.
* Subject is known to have tested positive for human immunodeficiency virus (HIV).
* Subject has a clinically significant abnormality on screening evaluation including physical examination, vital signs, ECG, or laboratory tests that the investigator in consultation with the medical monitor considers to be inappropriate to allow participation in the study.
* The subject's screening ECG shows a corrected QT interval using Fridericia's formula (QTcF) of ≥ 450 msec for male subjects or ≥ 470 msec for female subjects.
* The subject's screening hematology results show an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value ≥ 2 times the upper limit of normal (ULN), or a blood urea nitrogen (BUN) value ≥ 1.5 times the ULN for the reference lab.
* Subject who is currently participating or has participated in a clinical trial within the last 180 days or who participated in more than 2 clinical trials within the past year. This includes studies using marketed compounds or devices.
* Subject is at high risk of non-compliance in the investigator's opinion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 341 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (31):
- United States (31):
  - Pharmacology Research Institute, Encino, California
  - Collaborative Neuroscience Network Inc, Garden Grove, California
  - University of California at Irvine, Irvine, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Excell Research, Inc, Oceanside, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Clinical Neuroscience Solutions Inc., Jacksonville, Florida
  - Florida Research Center, Maitland, Florida
  - Miami Research Associates, Miami, Florida
  - Research Centers of America, LLC, Oakland Park, Florida
  - Medical Research Group of Central Florida, Sanford, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Goldpoint Clinical Research, Indianapolis, Indiana
  - IPS Research Company, Oklahoma City, Indiana
  - Rochester Center for Behavioral Health, Rochester Hills, Michigan
  - Midwest Research Group, Saint Charles, Missouri
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Brooklyn Medical Institutes, LLC, Brooklyn, New York
  - Duke Child and Family Study Center, Durham, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - CRI Lifetree, Philadelphia, Pennsylvania
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - Future Search Clinical Trials, LP, Austine, Texas
  - NeuroScience, Inc, Herndon, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington
  - Summit Research Network, LLC-Seattle, Seattle, Washington

REFERENCES:
- [Derived] Hopkins SC, Sunkaraneni S, Skende E, Hing J, Passarell JA, Loebel A, Koblan KS. Pharmacokinetics and Exposure-Response Relationships of Dasotraline in the Treatment of Attention-Deficit/Hyperactivity Disorder in Adults. Clin Drug Investig. 2016 Feb;36(2):137-46. doi: 10.1007/s40261-015-0358-7. PMID 26597180

RESULTS

PARTICIPANT FLOW:
Groups:
- SEP-225289 4mg: SEP-225289 4mg once daily taken as a combination of SEP-225289 2mg and placebo capsules to achieve 4mg QD doses
  SEP-225289: SEP-225289 4mg once daily
  SEP-225289: SEP-225289 8mg once daily
- SEP-225289 8mg: SEP-225289 8mg once daily taken as a combination of SEP-225289 2mg and placebo to achieve 8mg QD doses
  SEP-225289: SEP-225289 4mg once daily
  SEP-225289: SEP-225289 8mg once daily
Period: Overall Study
Arm/Group | SEP-225289 4mg | SEP-225289 8mg | Placebo
Started | 116 | 115 | 110
Completed | 96 | 59 | 100
Not Completed | 20 | 56 | 10
Not completed — Adverse Event | 12 | 32 | 2
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Lost to Follow-up | 2 | 7 | 1
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 2
Not completed — Non-complance with study drug | 0 | 4 | 1
Not completed — Non-compliant with study visits | 0 | 0 | 1
Not completed — SAE not related to study drug | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 10 | 3

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | SEP-225289 4mg | SEP-225289 8mg | Placebo | Total
Number analyzed (Participants) | 114 | 107 | 110 | 331
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 114 | 107 | 110 | 331
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.2 (10.06) | 34.5 (11.15) | 33.9 (11.03) | 34.2 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 43 | 44 | 137
  Male | 64 | 64 | 66 | 194
Region of Enrollment [Number; unit: participants]
  United States | 114 | 107 | 110 | 331

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 4 in ADHD Symptoms Measured With the ADHD Rating Scale Version IV With Adult Prompts (ADHD RS IV)
Description: The ADHD RS-IV with adult prompts is an 18 item scale based on the DSM IV TR criteria for ADHD that provides a rating of the severity symptoms. Scoring is based on a 4 point Likert-type severity scale where 0 = none, 1 = mild, 2 = moderate, and 3 = severe. Clinicians scored the highest score that was generated for the prompts for each item. The ADHD rating scale total score is defined as sum of all 18 item scale scores.
Time Frame: 4 Weeks
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SEP-225289 4mg | SEP-225289 8mg | Placebo
Number analyzed (Participants) | 114 | 107 | 110
units on a scale | -12.38 (1.07) | -13.88 (1.20) | -9.7 (1.07)
Statistical Analysis 1: Comparison: Placebo; The 4 mg and 8 mg SEP 225289 groups were compared to placebo using a MMRM analysis. The MMRM model included treatment, visit (as a categorical variable), pooled center, baseline ADHD RS-IV with adult prompts score, and treatment-by-visit interaction. An unstructured covariance matrix was used for the within subject correlation; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -9.7
Statistical Analysis 2: Comparison: SEP-225289 4mg; The 4 mg SEP 225289 group was compared to placebo using a MMRM analysis. The MMRM model included treatment, visit (as a categorical variable), pooled center, baseline ADHD RS-IV with adult prompts score, and treatment-by-visit interaction. An unstructured covariance matrix was used for the within subject correlation; Test type: Superiority or Other; p = 0.076, Mixed Models Analysis; P-values of SEP 225289 4 mg versus placebo at Week 4 was adjusted for multiple comparisons using the Hochberg procedure; Mean Difference (Final Values) = -12.38
Statistical Analysis 3: Comparison: SEP-225289 8mg; The 8 mg SEP 225289 group was compared to placebo using a MMRM analysis. The MMRM model included treatment, visit (as a categorical variable), pooled center, baseline ADHD RS-IV with adult prompts score, and treatment-by-visit interaction. An unstructured covariance matrix was used for the within subject correlation; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis — p-value of SEP 225289 8 mg versus placebo at Week 4 was adjusted for multiple comparisons using the Hochberg procedure; Mean Difference (Final Values) = -13.88

2. Secondary Outcome: Change From Baseline in ADHD Symptoms Measured With the ADHD RS IV at Weeks 1, 2, 3.
Description: The ADHD RS-IV with adult prompts is an 18 item scale based on the DSM IV TR criteria for ADHD that provides a rating of the severity symptoms. Scoring is based on a 4 point Likert-type severity scale where 0 = none, 1 = mild, 2 = moderate, and 3 = severe. Clinicians scored the highest score that was generated for the prompts for each item. The ADHD rating scale total score is defined as sum of all 18 item scale scores (range 0 - 54).
Time Frame: Weeks 1, 2, 3
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SEP-225289 4mg | SEP-225289 8mg | Placebo
Number analyzed (Participants) | 116 | 107 | 110
units on a scale
  Week 1 | -7.46 (0.77) | -7.83 (0.8) | -7.88 (0.79)
  Week 2 | -10.09 (0.91) | -11.03 (0.97) | -9.14 (0.92)
  Week 3 | -12.16 (0.99) | -12.79 (1.09) | -9.62 (1.0)

3. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity of Illness Scale (CGI S) at Weeks 1, 2, 3, 4.
Description: The CGI-S modified asked the clinician one question: Considering your total clinical experience with adult ADHD, how mentally ill is the subject at this time?".The clinician's answer was rated on the following 7-point scale: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = ng the most extremely ill subjects.
Time Frame: Weeks 1, 2, 3, 4
Population: Intent to treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SEP-225289 4mg | SEP-225289 8mg | Placebo
Number analyzed (Participants) | 116 | 107 | 110
units on a scale
  Week 1 | -0.44 (0.066) | -0.43 (0.069) | -0.45 (0.067)
  Week 2 | -0.74 (0.085) | -0.74 (0.091) | -0.61 (0.086)
  Week 3 | -0.98 (0.091) | -0.93 (0.102) | -0.69 (0.092)
  Week 4 | -1.08 (0.103) | -1.14 (0.118) | -0.74 (0.103)

4. Secondary Outcome: Change From Baseline in the Inattentiveness and Hyperactivity Subscales of the ADHD RS IV at Weeks 1, 2, 3, 4
Description: The ADHD RS-IV with adult prompts is an 18 item scale based on the DSM IV TR criteria for ADHD that provides a rating of the severity symptoms. Scoring is based on a 4 point Likert-type severity scale where 0 = none, 1 = mild, 2 = moderate, and 3 = severe. Clinicians scored the highest score that was generated for the prompts for each item. The even number items (2, 4, 6, 8, 10, 12, 14, 16, 18) assess hyperactive impulsive symptoms and the odd number items (1, 3, 5, 7, 9, 11, 13, 15, 17) assess inattentive symptoms. The ADHD inattentiveness subscale score is defined as sum of items (1, 3, 5, 7, 9, 11, 13, 15, 17) scores (range 0 - 27). The ADHD hyperactive impulsive subscale score is defined as sum of items (2, 4, 6, 8, 10, 12, 14, 16, 18) scores (range 0 - 27).
Time Frame: Weeks 1, 2, 3, 4
Population: Intent to treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SEP-225289 4mg | SEP-225289 8mg | Placebo
Number analyzed (Participants) | 116 | 107 | 110
units on a scale
  inattentivenes Week 1 | -4.23 (0.465) | -4.61 (0.483) | -4.64 (0.474)
  inattentivenes Week 2 | -5.75 (0.539) | -6.32 (0.581) | -5.43 (0.546)
  inattentivenes Week 3 | -6.93 (0.60) | -7.03 (0.669) | -5.89 (0.606)
  inattentivenes Week 4 | -7.0 (0.641) | -7.97 (0.732) | -5.61 (0.643)
  hyperactivity Week 1 | -3.23 (0.391) | -3.20 (0.405) | -3.26 (0.399)
  hyperactivity Week 2 | -4.35 (0.462) | -4.71 (0.498) | -3.75 (0.467)
  hyperactivity Week 3 | -5.23 (0.496) | -4.78 (0.553) | -3.78 (0.501)
  hyperactivity Week 4 | -5.39 (0.536) | -5.94 (0.615) | -4.13 (0.536)

5. Secondary Outcome: The Number of Responders at Weeks 1, 2, 3, 4. A Responder is Defined as a Subject With a ≥ 30% Improvement in ADHD Symptoms Compared With Baseline as Measured by the ADHD RS IV.
Time Frame: Weeks 1, 2, 3, 4
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | SEP-225289 4mg | SEP-225289 8mg | Placebo
Number analyzed (Participants) | 116 | 107 | 110
participants
  Week 1 | 36 | 35 | 35
  Week 2 | 44 | 39 | 39
  Week 3 | 55 | 43 | 36
  Week 4 | 49 | 38 | 40

6. Secondary Outcome: Change From Baseline in the Wender-Reimher Adult Attention Deficit Disorder Scale (WRAADDS) as Measured at Weeks 1, 2, 3, 4.
Description: The WRAADDS measured the severity of the target symptoms of adults with ADHD. It measured symptoms in 7 categories: attention difficulties, hyperactivity/restlessness, temper, affective lability, emotional overreactivity, disorganization, and impulsivity. The scale rated individual items from 0 to 2 (0 = not present, 1 = mild, 2 = clearly present) and summarized each of the 7 categories on a 0 to 4 scale (0 = none, 1 = mild, 2 = moderate, 3 = quite a bit, 4 = very much). The WRAADDS total score is defined as sum of all 28 item subscores (range 0 - 56).
Time Frame: Weeks 1, 2, 3, 4
Population: Intent to treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SEP-225289 4mg | SEP-225289 8mg | Placebo
Number analyzed (Participants) | 116 | 107 | 110
units on a scale
  Week 1 | -5.9 (0.783) | -6.97 (0.813) | -6.87 (0.80)
  Week 2 | -8.85 (0.919) | -9.11 (0.992) | -8.10 (0.933)
  Week 3 | -10.74 (0.957) | -9.84 (1.07) | -8.15 (0.967)
  Week 4 | -11.02 (1.005) | -11.91 (1.166) | -8.97 (1.004)

ADVERSE EVENTS:
Time Frame: From baseline to week 4 for double-blind treatment, then 2 weeks of follow-up
Arm/Group | SEP-225289 4mg | SEP-225289 8mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/116 | 1/111 | 0/110
Other Adverse Events (participants affected / at risk) | 88/116 | 89/111 | 65/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEP-225289 4mg (N=116) | SEP-225289 8mg (N=111) | Placebo (N=110)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemi (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEP-225289 4mg (N=116) | SEP-225289 8mg (N=111) | Placebo (N=110)
Combined insomniaa (Psychiatric disorders) | 40 (45) | 50 (55) | 17 (18)
Insomnia (Psychiatric disorders) | 29 (32) | 41 (46) | 11 (12)
Anxiety (Psychiatric disorders) | 11 (11) | 10 (11) | 2 (2)
Initial insomnia (Psychiatric disorders) | 4 (5) | 6 (6) | 3 (3)
Middle insomnia (Psychiatric disorders) | 4 (4) | 5 (5) | 2 (2)
Depressed mood (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 2 (2) | 2 (2) | 5 (5)
Panic attack (Psychiatric disorders) | 0 (0) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 15 (19) | 12 (12) | 12 (16)
Dizziness (Nervous system disorders) | 8 (8) | 9 (9) | 1 (1)
Tension headache (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 9 (9) | 19 (19) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (7) | 11 (11) | 3 (6)
Irritability (General disorders) | 10 (10) | 10 (10) | 9 (9)
Fatigue (Gastrointestinal disorders) | 7 (9) | 8 (8) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12) | 25 (26) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (3) | 6 (6)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 3 (3)
Weight decreased (Investigations) | 3 (4) | 6 (6) | 1 (1)
Palpitations (Cardiac disorders) | 6 (6) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS agreement between Principal Investigator and Sponsor that restricts PI's rights to discuss or publish trial results after trial is completed.

In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication provided, if a multicenter publication is not forthcoming within 24 months post completion of study at all sites, PI shall be free to publish.